CLINICAL TRIAL: NCT05159089
Title: A Socio-ecological Approach to Reduce the Physical Activity Drop-out Ratio in Primary Care-based Patients With Type 2 Diabetes: The SENWI Study Protocol for a Randomized Control Trial.
Brief Title: Physical Activity Drop-out Ratio in Patients Living With Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Vic - Central University of Catalonia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Uvicucc
Record Dates: First submitted 2021-11-02; First posted 2021-12-15 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Diabetes Mellitus, Type 2; Adherence, Patient; Physical Inactivity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Patient Compliance; Sedentary Behavior | interventions — Nordic Walking

STUDY DESIGN:
Intervention Model Description: A mixed methods research model will be used. A prospective and longitudinal three-arm randomized control trial with blinded evaluators will be needed to compare the efficacy of the interventions. Outcomes will be assessed at baseline, month three (end of intervention), and at months 12 and 24 (9 and 21-month post-intervention), which will be the main outcome assessment. The study protocol has been developed based on the Standard Protocol Items: Recommendation for Interventional Trials (SPIRIT) guidelines. On the other hand, a qualitative analysis using semi-structural interviews should help to understand both the reasons for the (un)efficacy and the patients' and HCP's perceptions about the intervention. Qualitative outcomes will be assessed at month three (end of intervention) and at month 24 (21-month post-intervention).
Who Masked: Investigator, Outcomes Assessor
Masking Description: The trial has an open design with a blind assessment of outcomes. Researchers conduction the baseline assessments will be blind to group allocation. The statistician (RMV) will also be blind to group allocation until the completion of the statistical analysis. Participants will be asked not to reveal group allocation when undergoing follow-up measurements. To assess the extent to which blinding has been preserved, researchers will record the number of cases in which allocation was revealed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nordic Walking Group (Active Comparator): Each group will be received 26 sessions of nordic walking. In each session, the intensity will be controlled and expected to be between 3 to 5 in the Borg scale adaptation. Patients will receive a schedule with all three-month sessions.
  Interventions: Behavioral: Nordic Walking
- Physical activity base on SEM (Socioecological models) (Experimental): The intervention group based on SEM will apply nordic walking in the same way as the Nordic Walking group. However, in this group, instructors will apply a SEM (instructors will not be the same as in the Nordic Walking group): in each session, the instructors in charge of the Nordic Walking will be also in charge to prescribe the PA.
  Interventions: Behavioral: Socioecological model apply to reduce physical activity drop out in type 2 diabetes patients
- Congrol group (No Intervention): Control group outcomes assessment will be the same as the intervention group. However, they will receive common health care professional advice. A common health care professional advice used to recommend patients to walk more and do more PA or physical exercise at the gym. Visits with doctors and nurses will be the same as the intervention group. The difference will be that at intervention group nurses will refer participants to the instructor's physiotherapist to promote PA throughout nordic walking and use the SEM to apply it.

INTERVENTIONS:
Behavioral: Socioecological model apply to reduce physical activity drop out in type 2 diabetes patients — To implement this model this intervention aims to address three key elements: 1) prepare the user; 2) structure the action; and 3) design the context.
  These goals will be worked in each session of Nordic Walking during the warm-up and cool-down and, if necessary, during the session (as long as it's non-stop or slowing down).
  Arms: Physical activity base on SEM (Socioecological models)
Behavioral: Nordic Walking — Sessions will be progressive: the first month will long 30 minutes, the second month 35 minutes, and the third month 40 minutes (without 10 minutes warm-up and 10 minutes cool-down each session). The track will not have more than 100 accumulate high and will allow doing 5 kilometers without stopping. The meeting point will be between the Biomedical Research Park (Barcelona) and Hospital del Mar (nearby CAP Sant Joan). All sessions will be conducted by an instructor of nordic walking physiotherapists.
  Arms: Nordic Walking Group

SUMMARY:
Physical activity (PA) - understood as any bodily movement produced by skeletal muscular that requires energy expenditure, related to leisure time, for transport to get to and from places, or part of a person's work - is a powerful force for good regarding type 2 diabetes mellitus (T2DM). However, fewer T2DM patients sustain the lifestyle recommendations suggested by health care professionals (HCP): 40% of patients did not follow-up on general medical recommendations regarding lifestyle changes. Using a socio-ecological approach - that aims to deal with the different levels of PA influences - may be a good solution to integrate the behaviour change techniques in health care professionals' consultations to prescribe PA efficiently.

The investigators' protocol has two aims. The primary aim is to evaluate the effectiveness of theory-driven PA intervention based on SEM among people living with T2DM. A secondary aim is to explore the feasibility and perceptions/experiences on the PA adherence process in T2DM patients while using the socio-ecological approach and to understand the HCP's viewpoint in its applicability in the Spanish Healthcare system. The investigators want to know the how, not the what, related to PA prescription.

DETAILED DESCRIPTION:
Physical activity (PA) - understood as any bodily movement produced by skeletal muscles that require energy expenditure, related to leisure time, for transport to get to and from places, or part of a person's work - is a powerful force for good regarding type 2 diabetes mellitus (T2DM). A recent meta-analysis has confirmed a positive dose-response relationship between markers of glucose control and increasing daily PA (a 20% increase in adherence or two sessions/month was associated with a 0.15% - 2 mmol/mol - decrease in HbA1c). Adhering to regular PA - understood as not dropping out the new PA behaviour adopted - is a way to control T2DM and promote people living with T2DM self-management. Still, fewer T2DM patients sustain the lifestyle recommendations suggested by health care professionals (HCP): 40% of patients did not follow up on general medical recommendations regarding lifestyle changes.

Socioeconomic status and health or social inequity, immediate and non-negotiable patients' needs and adherence skills rarely discussed by HCP, urban planning and political decisions about PA, or physical inactive workplaces may be reasons for these poor results in sustaining PA lifestyle recommendations.

Researchers have proposed aerobic or resistance exercise - understood as PA planned, structured, and realized during the leisure-time - like Nordic walking, high-intensity training, or lifting weights to increase PA levels throughout exercise among T2DM patients. Despite all options having good results in metabolic and patients' health outcomes, it seems that they are only used in well-controlled studies rather than in healthcare: that may be due to the HCP difficulty and lack of time, support, and knowledge to prescribe this type of aerobic and resistance exercise.

As a result, HCP most common prescription is based on walking, as it is easy to recommend and to do it by people living with T2DM without contraindications. However, only doing that recommendation will be not efficient nor effective to improve PA levels among people living with T2DM. For example, the more prevalent of people living with T2DM belongs to the lower-medium class, which usually live in neighborhoods with poor walkability and parks or green spaces. As a result, patients used to drop out in the long run and despite decades of this type of recommendation, PA population levels are still a problem to be faced. With that panorama, HCP may intentionally withdraw from PA prescriptions to protect patients who find it difficult to keep going.

In this context, ineffective primary-care-based PA prescription risks missing out on the health benefits of the powerful factors that manage people living with T2DM health-related outcomes. Moreover, ineffective primary-care-based PA prescription may enhance socioeconomic barriers and health inequity in these patients. Therefore, given the scale and span of these PA biological and social benefits, it remains a Public Health priority to deploy more effective ways to implement day-to-day PA life. Doing so will be helpful for health patients and for both HCP that used to have not enough time to prescribe exercise effectivity and Public Health expenses in T2DM patients.

Knowing the health need of PA, it is necessary to address PA prescription on how, where, when, and with whom to do it. In this sense, different behaviour changes techniques (BCTs) have been used to face the PA adherence issue and reduce the drop-out ratio: goal setting, action planning, problem solving or social support are a few examples of BCTs used. BCTs results seem hopeful; they improve PA adherence both in the short and in the long run.

However, despite these results, BCTs are still generally not used by HCPs to prescribe PA efferently. HCPs' lack of time and lack of institutional support, and also gathering bad patients' results discourage HCPs to keep trying to change people with T2DM behaviour about PA. Even more, BCTs are still focused on individual responsibility, usually forgetting all the sociocultural barriers as social inequity or poor urban planning. In this context, both HCP and people living with T2DM feel powerless in front of complex multi-component sociocultural situations. BTCs need to take into consideration these complex multicomponent socio-cultural situations to be applied efficiently by HCPs in real-world situations.

In this complex multicomponent sociocultural situation, using a socio-ecological approach - that aims to deal with the different levels of PA influences - may be a good solution to integrate the BCTs in HCPs consultations to prescribe PA efficiently. The socio-ecological model (SEM) considers the complex interplay between individual, relationship, community, and societal factors to influence personal behaviour. This approach focuses on integrating these different levels to change the physical and social environments rather than modifying only individual health behaviours. That may involve facing different sociocultural barriers as socioeconomic status and social inequity (e.g. delivering free PA with a specialist), gender and age discrimination (e.g. explaining to patients what PA is important too), or urban planning (e.g. HCPs should be shown to people living with T2DM some green spaces to do PA). Otherwise, the responsibility to deal with PA adherence will rely on powerless people living with T2DM and HCP alike.

Our protocol has two aims. The primary aim is to evaluate the effectiveness of theory-driven PA intervention based on a SEM among people living with T2DM. A secondary aim is to explore the feasibility and perceptions/experiences on the PA adherence process in T2DM patients while using the socio-ecological approach and to understand the HCP's viewpoint in its applicability in the Spanish Healthcare system. The investigators want to know the how, not the what, related to PA prescription.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with T2D
2. Be eligible to be referred by their doctors for PA intervention;
3. Have no major physical limitations prescribed by the doctor or any HCP
4. Physical inactive according to the General Practice Physical Activity Questionnaire - GPPAQ screening tool.

Exclusion Criteria:

1. Pregnant patients or have T2D due to gestation
2. Inability to freely consent to take part in the study
3. Inability to understand the study materials or PA intervention
4. T2D patients with complications as neuropathy, retinopathy, and nephropathy
5. Contraindications to do PA
6. Body Mass Index over 34,9

Ages: 45 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Participant physical activity drop-out ratio | up to 12 weeks
  During the intervention, drop out will be considered as less than 80% of assistance at schedule sessions.
  After the intervention, PA drop out will be measured asking the participants if they continue to undertake PA in their daily life. Participants will be asked once a month until the 24-month (21-month post-intervention) throughout telephone calls and messages (using ecological memorial assessments) about the following-up. What will be important if they do any kind of PA, no matter what kind. The answer will be registered as yes or no.
Participant physical activity levels | up to 12 weeks
  PA levels will be assessed throughout activPAL3™ micro
Participant physical activity levels | 2 years
  PA levels will be assessed throughout activPAL3™ micro
Metabolic participants outcomes | up to 12 weeks
  HbA1c analysis from blood sample
Metabolic participants outcomes | 2 years
  HbA1c analysis from blood sample

SECONDARY OUTCOMES:
Socioeconomic participant status | Before the intervention
  Socioeconomic status will be asses using three different levels: occupation, education level and annual income. All three levels will be combined to determine if participants belong to a high, medium or low socioeconomic status.

OTHER OUTCOMES:
Medication patients intake | up to 12 weeks
  This outcome will be assessed as a category outcome with three options: i) patients medication intake is reduced or ii) patients medication intake is the same or iii) patients medication intake is increased.
Medication patients intake | 2 years
  This outcome will be assessed as a category outcome with three options: i) patients medication intake is reduced or ii) patients medication intake is the same or iii) patients medication intake is increased.

CONTACTS AND LOCATIONS:
Overall Officials: Guillem Jabardo-Camprubí, Principal Investigator — University of Vic - Central University of Catalonia
Locations (5):
- Spain (5):
  - Hospital Sant Bernabé, Berga, Barcelona
  - Centre d'Atenció Primaria Anoia, Igualada, Barcelona
  - Centre d'Atenció Primaria les Bases, Manresa, Barcelona
  - Monistrol de Montserrat CAP, Monistrol de Montserrat, Barcelona
  - Centre d'Atenció Primaria Vic Sud, Vic, Barcelona

IPD SHARING:
Plan to Share IPD: No
Publishing an article in an open journal

REFERENCES:
- [Background] Jabardo-Camprubi G, Donat-Roca R, Sitja-Rabert M, Mila-Villarroel R, Bort-Roig J. Drop-out ratio between moderate to high-intensity physical exercise treatment by patients with, or at risk of, type 2 diabetes mellitus: A systematic review and meta-analysis. Physiol Behav. 2020 Mar 1;215:112786. doi: 10.1016/j.physbeh.2019.112786. Epub 2019 Dec 18. PMID 31863856
- [Derived] Jabardo-Camprubi G, Bort-Roig J, Donat-Roca R, Mila-Villarroel R, Sitja-Rabert M, McKenna J, Puig-Ribera A. A socio-ecological approach to reduce the physical activity drop-out ratio in primary care-based patients with type 2 diabetes: the SENWI study protocol for a randomized control trial. Trials. 2022 Oct 3;23(1):842. doi: 10.1186/s13063-022-06742-7. PMID 36192800